CLINICAL TRIAL: NCT06054464
Title: A Phase 1, Open-Label, Non-Randomized, Two-Part, Fixed-Sequence, Study to Evaluate the Effects of Acid Reducing Agents on the Pharmacokinetics of PC14586 in Healthy Volunteers
Brief Title: A Study to Investigate the Effects of Acid Reducing Agents on Pharmacokinetics of PC14586 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PMV Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PMV-586-104
Record Dates: First submitted 2023-09-08; First posted 2023-09-26 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Y220C; PC14586; PMV Pharma; PMV; Acid Reducing Agent; p53; DDI; Phase 1; p53 mutation; TP53 mutation; TP53; p53 mutant; p53 reactivator
MeSH Terms: interventions — Rabeprazole; Famotidine

STUDY DESIGN:
Intervention Model Description: The treatment duration will be up to: 1 day for Treatment Period 1 (PC14586) and 4 days for Treatment Period 2 (PC14586 + ARA) for Parts 1 and 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: PC14586 and rabeprazole (Experimental): Healthy participants will receive a single, oral dose of PC14586 on day 1. On days 11-13, participants will receive an oral daily dose of rabeprazole. On day 14, participants will receive a co-administration dose of rabeprazole and PC14586. Rabeprazole will be given 1 hour prior to PC14586. Participants will be given a low-fat meal 30 minutes prior to PC14586 dosing.
  Interventions: Drug: PC14586; Drug: Rabeprazole
- Part 2: PC14586 and famotidine (Experimental): Healthy participants will receive a single, oral dose of PC14586 on day 1. On days 11-13, participants will receive a twice daily, oral dose of famotidine. On day 14, participants will receive PC14586 two hours before a dose of famotidine. Participants will be given a low-fat meal 30 minutes prior to PC14586 dosing.
  Interventions: Drug: PC14586; Drug: Famotidine

INTERVENTIONS:
Drug: PC14586 — Part 1 and Part 2: Single, oral dose of PC14586 on day 1 and single, oral dose of PC14586 on day 14.
Drug: Rabeprazole — Part 1: Daily oral dose of rabeprazole on days 11-14.
  Arms: Part 1: PC14586 and rabeprazole
Drug: Famotidine — Part 2: Twice daily oral dose of famotidine on days 11-13. Single, oral dose of famotidine on day 14.
  Arms: Part 2: PC14586 and famotidine

SUMMARY:
This study will assess the effect of a Proton Pump Inhibitor (PPI) (rabeprazole) on the pharmacokinetics (PK) of PC14586 and the effect of an H2-receptor antagonist (famotidine) on the PK of PC14586

DETAILED DESCRIPTION:
PC14586 is a first-in-class, oral, small molecule p53 reactivator that is selective for the TP53 Y220C mutation. This study will investigate the effects of acid reducing agents on the pharmacokinetics of PC14586.

This is a 2-part, open-label, two-period, fixed-sequence study in healthy participants with each participant used as his/her own control to assess the effect of rabeprazole (Part 1) or famotidine (Part 2) on the PK of PC14586. The results from Part 1 will be analyzed before deciding to, if applicable, progress to Part 2. Part 2 of the study will only be initiated if the findings from Part 1 show an interaction or are inconclusive.

Approximately 25 participants will be enrolled in Part 1 and approximately 25 participants will be enrolled in Part 2. The Study timelines reflect both Part 1 and Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking males and females, 18-55 years of age, with BMI between 18.5 - 30 kg/m2 inclusive.
2. Agree to use a highly effective method of contraception from 14 days before check-in through 90 days after last dose of study drug.
3. Participants who are capable of giving signed informed consent.

Exclusion Criteria:

1. Participants with significant history or clinical manifestation of any medical condition, disease or disorder, as determined by the Investigator.
2. Positive hepatitis panel and/or positive human immunodeficiency virus test.
3. Use or intend to use any prescription and/or nonprescription medications/products within 14 days prior to check-in.
4. Participation in a clinical study involving last administration of an investigational drug within the past 30 days prior to screening.
5. Participant has blood pressure > 140 mm systolic or > 90 mm diastolic at Screening or Day - 1.
6. Participants with a germline TP53 Y220C mutation at Screening.
7. Participant has smoked or used other nicotine-containing products (snuff, chewing tobacco, cigars, pipes, vaporizer, or nicotine-replacement products such as nicotine chewing gum and nicotine plasters) during the 3 months before the Screening Visit.
8. Participant has history of alcohol and/or illicit drug abuse within 5 years of Screening.
9. Participant is unwilling to avoid use of alcohol or alcohol-containing foods, medications, or beverages, 48 hours prior to admission until discharge from the study center.
10. Participant has a history of hypersensitivity to the study drug (PC14586), rabeprazole (Part 1), or famotidine (Part 2) or any of the excipients or to medicinal products with similar chemical structures.
11. Female participant that is breastfeeding (or bottle feeding with their breast milk) or female participant with a positive serum pregnancy test at the Screening Visit or positive serum or urine pregnancy test at Day -1 (admission).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Characterize the Maximum Plasma Concentration (Cmax) of PC14586 when co-administered with rabeprazole. | 20 days
  Determine the Cmax of PC14586 when co-administered with rabeprazole in plasma.
Part 1: Characterize the total drug exposure to the last measurable concentration (AUC0-last) of PC14586 when co-administered with rabeprazole. | 20 days
  Determine the AUC0-last of PC14586 when co-administered with rabeprazole in plasma.
Part 1: Characterize the total drug exposure (AUC0-inf) of PC14586 when co-administered with rabeprazole. | 20 days
  Determine the AUC0-inf of PC14586 when co-administered with rabeprazole in plasma.
Part 1: Characterize the time to peak drug concentration (Tmax) of PC14586 when co-administered with rabeprazole. | 20 days
  Determine the Tmax of PC14586 when co-administered with rabeprazole in plasma.
Part 2: Characterize the Maximum Plasma Concentration (Cmax) of PC14586 when co-administered with famotidine. | 20 days
  Determine the Cmax of PC14586 when co-administered with famotidine in plasma.
Part 2: Characterize the total drug exposure to the last measurable concentration (AUC0-last) of PC14586 when co-administered with famotidine. | 20 days
  Determine the AUC0-last of PC14586 when co-administered with famotidine in plasma.
Part 2: Characterize the total drug exposure (AUC0-inf) of PC14586 when co-administered with famotidine. | 20 days
  Determine the AUC0-inf of PC14586 when co-administered with famotidine in plasma.
Part 2: Characterize the time to peak drug concentration (Tmax) of PC14586 when co-administered with famotidine. | 20 days
  Determine the Tmax of PC14586 when co-administered with famotidine in plasma.

SECONDARY OUTCOMES:
Part 1: Characterize the total drug exposure from time zero to 24 hours (AUC0-24) for PC14586 when co-administered with rabeprazole. | 20 days
  Determine the AUC0-24 of PC14586 when co-administered with rabeprazole in plasma.
Part 1: Characterize the total drug exposure from time zero to 96 hours (AUC0-96) for PC14586 when co-administered rabeprazole. | 20 days
  Determine the AUC0-96 of PC14586 when co-administered with rabeprazole in plasma.
Part 1: Characterize the percent AUCinf due to extrapolation beyond tlast (AUC%extrap) for PC14586 when co-administered with rabeprazole. | 20 days
  Determine the AUC%extrap of PC14586 when co-administered with rabeprazole in plasma.
Part 1: Characterize the half-life (t1/2) for PC14586 when co-administered with rabeprazole. | 20 days
  Determine the t1/2 of PC14586 when co-administered with rabeprazole in plasma.
Part 1: Characterize the clearance (CL/F) for PC14586 when co-administered orally with rabeprazole. | 20 days
  Determine the CL/F of PC14586 when co-administered orally with rabeprazole in plasma.
Part 1: Characterize the volume of distribution (Vz/F) for PC14586 when co-administered orally with rabeprazole. | 20 days
  Determine the Vz/F of PC14586 when co-administered orally with rabeprazole in plasma.
Part 1: Characterize the apparent terminal elimination rate (lambda Z) for PC14586 when co-administered orally with rabeprazole. | 20 days
  Determine the lambda Z of PC14586 when co-administered orally with rabeprazole in plasma.
Part 1: Identification of the Incidence of treatment emergent adverse events (TEAE) for PC14586 alone or when co-administered with rabeprazole. | 20 days
  Identify the incidence of TEAEs of PC14586 alone or when co-administered orally with rabeprazole in plasma.
Part 1: Identification of vital sign abnormalities after administration of PC14586 alone or when co-administered with rabeprazole. | 20 days
  Number of participants with abnormal vital signs.
Part 1: Identification of 12-lead electrocardiogram (ECG) abnormalities after administration of PC14586 alone or when co-administered with rabeprazole. | 20 days
  Number of participants with abnormal ECG results.
Part 1: Identification of laboratory abnormalities based on hematology and clinical chemistry after administration of PC14586 alone or when co-administered with rabeprazole. | 20 days
  Number of participants with an incidence of laboratory abnormalities in test results.
Part 2: Characterize the total drug exposure from time zero to 24 hours (AUC0-24) for PC14586 when co-administered with famotidine. | 20 days
  Determine the AUC0-24 of PC14586 when co-administered with famotidine in plasma.
Part 2: Characterize the total drug exposure from time zero to 96 hours (AUC0-96) for PC14586 when co-administered with famotidine. | 20 days
  Determine the AUC0-96 of PC14586 when co-administered with famotidine in plasma.
Part 2: Characterize the percent AUCinf due to extrapolation beyond tlast (AUC%extrap) for PC14586 when co-administered with famotidine. | 20 days
  Determine the AUC%extrap of PC14586 when co-administered with famotidine in plasma.
Part 2: Characterize the half-life (t1/2) for PC14586 when co-administered with famotidine. | 20 days
  Determine the t1/2 of PC14586 when co-administered with famotidine in plasma.
Part 2: Characterize the clearance (CL/F) for PC14586 when co-administered orally with famotidine. | 20 days
  Determine the CL/F of PC14586 when co-administered orally with famotidine in plasma.
Part 2: Characterize the volume of distribution (Vz/F) for PC14586 when co-administered orally with famotidine. | 20 days
  Determine the Vz/F of PC14586 when co-administered orally with famotidine in plasma.
Part 2: Characterize the apparent terminal elimination rate (lambda Z) for PC14586 when co-administered orally with famotidine. | 20 days
  Determine the lambda Z of PC14586 when co-administered orally with famotidine in plasma.
Part 2: Identification of the Incidence of treatment emergent adverse events (TEAE) for PC14586 alone or when co-administered with famotidine. | 20 days
  Identify the incidence of TEAEs of PC14586 alone or when co-administered orally with famotidine in plasma.
Part 2: Identification of vital sign abnormalities after administration of PC14586 alone or when co-administered with famotidine. | 20 days
  Number of participants with abnormal vital signs.
Part 2: Identification of 12-lead electrocardiogram (ECG) abnormalities after administration of PC14586 alone or when co-administered with famotidine. | 20 days
  Number of participants with abnormal ECG results.
Part 2: Identification of laboratory abnormalities based on hematology and clinical chemistry after administration of PC14586 alone or when co-administered with famotidine. | 20 days
  Number of participants with an incidence of laboratory abnormalities in test results.

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No